CLINICAL TRIAL: NCT01926470
Title: The Incidence of the Intravascular Injection During S1 Transforaminal Epidural Steroid Injection in Two Approaches: Anteroposterior Versus Oblique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 4-2013-0310
Record Dates: First submitted 2013-07-17; First posted 2013-08-21 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Lumbosacral Radicular Pain
Keywords: epidural injections, intravascular injection

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anteroposterior approach group (Experimental): anteroposterior approach group
  Interventions: Procedure: anteroposterior approach group
- oblique approach group (Active Comparator): oblique approach group
  Interventions: Procedure: oblique approach group

INTERVENTIONS:
Procedure: anteroposterior approach group — anteroposterior approach group (n=104): check intravascular injection while performing S1 transforaminal epidural steroid injection in anteroposterior view under fluoroscopy
  Arms: anteroposterior approach group
Procedure: oblique approach group — oblique approach group (n=104): same as anteroposterior approach group except using oblique view
  Arms: oblique approach group

SUMMARY:
Lumbosacral transforaminal epidural steroid injection (TFESI) is helpful for the treatment of lumbosacral radicular pain, but in case of intravascular injection, infrequently serious complication can be developed. Against this backdrop, if there is any difference of frequency of intravascular injection incidence during S1 TFESI between method in anteroposterior view and method in oblique view using Scotty dog, the result can be crucial factor in selecting the approach. In addition, appropriate volume of injection will be checked in each approach.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (20-80 years of age) who were scheduled to receive S1 transforaminal epidural steroid injection for lumbosacral radicular pain at our pain management clinic

Exclusion Criteria:

* pregnancy
* coagulopathy
* systemic infection
* any active infection at the injection site
* history of allergy to contrast media, local anesthetics, corticosteroid
* patients unable to communicate or patients with cognitive dysfunction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
the incidence of intravascular injection | 5 seconds after injection of contrast media via block needle.
  the incidence of intravascular injection in the anteroposterior approach group and the oblique approach group

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Al-Shaikh B, George William M, Van Zundert AA. Using atmospheric pressure to inflate the cuff of the Portex Laryngeal Mask. Anaesthesia. 2005 Mar;60(3):296-7. doi: 10.1111/j.1365-2044.2005.04135.x. No abstract available. PMID 15710025